CLINICAL TRIAL: NCT01631513
Title: An Open-label, Multi-center, Single-arm, Phase IV Clinical Trial Assessing Conversion From Hydrocodone, Oxycodone CR or Morphine SR to Tapentadol ER in Subjects With Moderate to Severe Chronic Low Back or OA Pain of the Hip or Knee
Brief Title: An Open-label Evaluation of Tapentadol Extended Release (ER) in Participants With Moderate to Severe Chronic Pain After Conversion From Hydrocodone, Oxycodone Controlled Release (CR), and/or Morphine Sustained Release (SR)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: It was a business decision to cancel this study in Aug. 2012.
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100757; R331333PAI4005 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2012-06-27; First posted 2012-06-29 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2016-11

CONDITIONS: Pain; Chronic Back Pain; Chronic Low Back Pain; Osteoarthritis Pain In The Hip or Knee
Keywords: Chronic Low Back Pain; Osteoarthritis Pain In The Hip or Knee; Oxycodone; Morphine, Hydrocodone; Tapentadol; NUCYNTA ER
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nucynta ER (Experimental): Nucynta ER will be 100 to 250 mg every 12 hours
  Interventions: Drug: Nucynta ER

INTERVENTIONS:
Drug: Nucynta ER — 100 to 250 mg every 12 hours
  Other Names: Nucynta Extended Release

SUMMARY:
The purpose of this study is to evaluate tapentadol Extended Release (ER) in the treatment of moderate to severe chronic pain in participants with a diagnosis of chronic low back pain (LBP) or osteoarthritis (OA) of the hip or knee after conversion from hydrocodone, oxycodone Controlled Release (CR), and/or morphine Sustained Release (SR).

DETAILED DESCRIPTION:
This is a multi-center, single group, open-label (all people know the identity of the intervention) treatment study to describe the overall clinical experience in participants with moderate to severe chronic low back pain or OA pain of the hip or knee, after conversion from hydrocodone, oxycodone CR, and/or morphine SR, using dose-conversion ratios of 1:5, 1:5 and 1:2.5, respectively.

Approximately 150 participants taking hydrocodone, oxycodone CR, and/or morphine SR with baseline pain intensity ≥4 (ie, pain intensity scores averaged over the last 4 days of the screening period on an 11-point numeric rating scale [NRS]) will be converted to an initial dose of tapentadol ER 100, 150 or 200 mg approximately every 12 hours based on their total daily dose of prior opioids. Enrollment of participants in any prior opioid group (hydrocodone, oxycodone CR, and/or morphine SR) may be stopped at any time during the study to ensure adequate representation of each prior opioid.

The study will consist of two periods: screening (1 Week) and treatment (4 weeks). The expected duration of participation for individual participants is approximately 5 weeks, including 4 weeks of active study treatment. The study will include scheduled visits and may also include unscheduled phone calls and site visits for dose adjustment and/or for safety evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of knee or hip osteoarthritis (OA) with history of pain at the reference joint or clinical diagnosis of low back pain (LBP) of non malignant origin for at least 3 months before the screening visit; Be taking hydrocodone, oxycodone CR, or morphine SR for the treatment of chronic LBP, or OA of the knee or hip for at least 2 weeks before the screening visit; Have a baseline pain intensity score of ≥4 on an 11-point pain intensity numeric rating scale; Be willing and able to independently communicate pain characteristics, complete all protocol required measurements/assessments without assistance, understand and complete self-administered questionnaires and adhere to the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Had surgery in the low back area or the reference joint within 3 months before the screening visit, or will not have fully recovered from surgery by the screening visit, or is expected to require surgical intervention in the low back area or the reference joint during participation in the study; For participants with OA of the hip or knee, has a clinical history and findings at the reference joint suggesting the pain is secondary to crystal-induced, metabolic, infectious, and/or autoimmune disease(s); Has a known history of severe chronic renal insufficiency, severely impaired hepatic function, or alanine aminotransferase or aspartate aminotransferase greater than three times the upper limit of normal; Has a history of seizure disorder, epilepsy, or recurrent seizures; Has any of the following within 1 year before the screening visit: mild/moderate traumatic brain injury, stroke, transient ischemic attack, or brain neoplasm; Has a known or suspected history of alcohol abuse in the past 10 years or any history of drug abuse; Has a history of malignancy within 2 years before the screening visit, with the exception of basal cell carcinoma that has been successfully treated; Has significant respiratory depression, acute or severe bronchial asthma, or hypercapnia and paralytic ileus; Has a known history of allergies, hypersensitivity, or contraindication to tapentadol, hydrocodone, morphine, oxycodone, or acetaminophen or their excipients; In a participant taking oxycodone CR or morphine SR at screening, is also taking more than 2 doses per day of an IR opioid for breakthrough pain (exclusion does not apply if prior opioid is hydrocodone); Is taking daily acetaminophen at a dose that exceeds 3,000 mg/day, including both acetaminophen and acetaminophen-containing combination products; Has received systemic corticosteroids within 4 weeks before the screening visit; For participant with OA, has received an injection of hyaluronic acid into the reference joint within 4 weeks before the screening visit; Has taken a monoamine oxidase inhibitor within 14 days before the screening visit; Has received an investigational drug or used an invasive investigational medical device within 30 days before the screening visit or is currently enrolled in an investigational study; Has previously participated in this clinical study; Is a woman who is pregnant, breast-feeding, or planning to become pregnant within 2 weeks after the last dose of study drug; Has any planned procedure that would require supplemental analgesics during the time of expected participation in the study; Has any significant pain condition other than chronic LBP or OA that, in the opinion of the investigator, could confound the assessment or self-evaluation of pain; Current diagnosis of fibromyalgia, complex regional pain syndrome, acute spinal cord compression, bowel or bladder dysfunction as a result of cauda equina compression, back pain caused by secondary infection, or pain caused by suspected neoplasm; Have answered "yes" to items 1 and 2 in the Columbia Suicide Severity Rating Scale administered at the screening visit.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2012-08 (Actual); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity from baseline to end of study as measured on an 11-point numeric rating scale (NRS) | Day 1 and Day 29
  The pain intensity NRS is a commonly used pain scale that is a core recommended outcome measure for chronic pain studies. A score of 0 indicates "no pain" and a score of 10 indicates "pain as bad as you can imagine." Change in pain intensity is measured from baseline to the end of treatment.

SECONDARY OUTCOMES:
11-point pain intensity numeric rating scale (NRS) (twice daily) and diary compliance | Day 1, Day 8, Day 15, Day 22, Day 29
  The pain intensity NRS is a commonly used pain scale that is a core recommended outcome measure for chronic pain studies. A score of 0 indicates "no pain" and a score of 10 indicates "pain as bad as you can imagine."
Quality of life as measured by the SF-12v2® Health Survey | Day 8, Day 15, Day 22, Day 29
  The SF-12v2® is a 12-item health survey instrument that is used to evaluate the subject's physical, social, and mental well-being. Results are expressed in terms of 2 composite scores: the Physical Component Scale (PCS) and the Mental Component Summary (MCS). PCS and MCS values can range from 0 to 100. Lowest scores mean very much below and highest scores mean very much above the general population average.
Pain interference as measured by the Brief Pain Intensity-Short Form (BPI-SF) questionnaire | Day 8, Day 15, Day 22, Day 29
  The BPI-SF is a self-administered, validated tool for the assessment of severity of pain and the impact of pain on daily functions, location of pain, pain medications, and amount of pain relief in the last week. The BPI-SF uses a numeric rating scale (NRS) from 0 to 10, lower score denotes less severity and impact, higher score denotes more severity and impact.
Sleep quality as measured by the Sleep Questionnaire | Day 1, Day 8, Day 15, Day 22, Day 29
  The 4-item Sleep Questionnaire is a validated instrument including the 4 main concepts that are considered standard and are consistently measured via sleep diaries: latency, time slept, number of awakenings, and quality experienced by the subject during the preceding night.
Extent of neuropathic pain as measured by the painDETECT questionnaire (PDQ) | Day 8, Day 29
  The PDQ is a simple evaluation tool to help identify the presence of neuropathic pain. It consists of 12 questions that ask about the intensity and quality of the patient's pain. A score between 0 and 12 is "negative" (no neuropathic pain component). A score between 19 and 38 is "positive" (presence of neuropathic component)". Scores from 13 to 18 are "unclear".
Participant rating of overall treatment status as measured by the patient global impression of change (PGIC) | Day 29
  The PGIC is a questionnaire that assesses the subject's global improvement since starting study treatment. It uses a 7-point NRS (1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (7):
- United States (7):
  - Jacksonville, Florida
  - Prairie Village, Kansas
  - Mandeville, Louisiana
  - Metairie, Louisiana
  - New Orleans, Louisiana
  - Oklahoma City, Oklahoma
  - Clinton, Utah